CLINICAL TRIAL: NCT04921163
Title: Children With Aluminium Contact Allergy: Oral Exposure Study (the Pancake Study)
Brief Title: Children With Aluminium Contact Allergy: Oral Exposure Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Allergy Research Center, Denmark (Other)
Responsible Party: Principal Investigator, Stine Hoffmann, MD, ph.d. student, National Allergy Research Center, Denmark
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-20060917
Record Dates: First submitted 2021-01-14; First posted 2021-06-10 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Contact Dermatitis; Contact Allergy; Aluminum Allergy
Keywords: vaccination granuloma; aluminium; contact allergy; exposure
MeSH Terms: conditions — Dermatitis, Contact; Dermatitis, Allergic Contact

STUDY DESIGN:
Intervention Model Description: double blinded cross over study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aluminium (Active Comparator): 4-day test periode with intake of aluminium pancakes
  Interventions: Dietary Supplement: sodium aluminium phospate (SALP)
- placebo (Placebo Comparator): 4-day test periode with aluminium-free pancakes
  Interventions: Dietary Supplement: Aluminium-free pancake
- second placebo (Placebo Comparator): Again a 4-day test periode with aluminium-free pancakes
  Interventions: Dietary Supplement: Aluminium-free pancake

INTERVENTIONS:
Dietary Supplement: sodium aluminium phospate (SALP) — 1 pancake daily for 4 days
  Arms: aluminium
Dietary Supplement: Aluminium-free pancake — 1 pancake daily for 4 days, without aluminium
  Arms: placebo; second placebo

SUMMARY:
Aluminium allergy is predominantly seen in children with small itchy nodules in the skin after vaccinations, so-called granulomas. We want to do an exposure study where aluminium allergic children have to eat aluminium pancakes for a short period of time. The purpose is to investigate whether a worsening of the children's symptoms can be detected, both itching of the granuloma, allergic rash on the skin and also the symptoms that are not measurable, such as headache, stomach ache and general agitation. We also want to examine the concentration of aluminium in the urine, which reflects the absorption of aluminum from the gastrointestinal tract.

DETAILED DESCRIPTION:
Parents of aluminium allergic children have reported that children may react with increased itching of their granulomas, skin symptoms in the form of redness, itching and rash, as well as symptoms such as headache, abdominal pain and agitation, by ingesting aluminium-containing foods.

Children are predominantly exposed to aluminium via the diet as they do not yet use aluminium-containing cosmetic products, stomach acid medicines or deodorants. The amount of aluminium in children's diet varies between 0.22-0.90 mg/kg body weight/week, depending on their age. In older children and adults, the intake is less related to the aluminium in infant formula, breakfast cereals and dried fruit, which is consumed more by children than adults.

With this study, we want to create an exposure study where children have to eat pancakes for a limited period of time, where aluminium has been used as baking soda, and for two control periods eat pancakes without aluminium.

Any symptoms occurring during periods could be used to investigate whether children with aluminium allergies generally react after intake of aluminium-containing foods and whether as such it is a consequential condition in some children or whether it is isolated cases. It is a very important issue to clarify with a view to proper advice, both with regard to the possible avoidance of specific foods and in the case of future vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* Children with contact allergies to aluminium, demonstrated by patch tests
* Activity (itching) of the granulom within the last six months
* Written consent obtained from all custodians

Exclusion Criteria:

* a detected food allergy for the remaining products in the pancakes (including wheat flour, eggs and milk)
* Children treated with topical and/or systemic steroid preparations during and up to 1 week before the start of the study.
* Children treated with systemic immune suppression during and up to 1 week before the start of the study.
* Children with kidney or bone disease.
* Children vaccinated during the study period
* Treatment with acid neutralising medicines during and up to 1 week before the start of the study
* Another reason for inability to cooperate, including lack of language skills in Danish or English in parents.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
granuloma | 1-7 days
  itch of existing granuloma evaluated on a Visual analogue scale 0-10
skin | 1-7 days
  flare-up of previous patch test area, evaluated on a visual scheme
subjective | 1-7 days
  headache, irritability, stomach ache evaluated on an adapted visual analogue scale 0-10

SECONDARY OUTCOMES:
sleep | 1-7 days
  disturbed sleep evaluated by an activity tracker watch during sleep. The watch records all movements during sleep, and we especially focus on the number of times the child wakes up at night

CONTACTS AND LOCATIONS:
Locations (1):
- National Allergy Research Centre, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No